CLINICAL TRIAL: NCT02200016
Title: Displacement of Popliteal Sciatic Nerve Catheters After Major Foot and Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Wulff Hauritz, Consultant, Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2014-000707-28
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain; Regional Anesthesia
Keywords: Postoperative pain; Regional anesteshia; Nerve catheters; Sciatic nerve catheters
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAX (Experimental): Ultrasound guided short axis (SAX) placement of sciatic nerve catheters
  Interventions: Procedure: Ultrasound guided short axis (SAX) placement of sciatic nerve catheters; Device: B Braun Contiplex S catheter
- LAX (Active Comparator): Ultrasound guided long axis (LAX) placement of sciatic nerve catheters
  Interventions: Procedure: Ultrasound guided long axis (LAX) placement of sciatic nerve catheters; Device: B Braun Contiplex S catheter

INTERVENTIONS:
Procedure: Ultrasound guided short axis (SAX) placement of sciatic nerve catheters — Sonosite EDGE ultrasound scanner guided insertion of a B Braun Contiplex S catheter along the short axis of the sciatic nerve behind the knee.
  Arms: SAX
Procedure: Ultrasound guided long axis (LAX) placement of sciatic nerve catheters — Sonosite EDGE ultrasound scanner guided insertion of a B Braun Contiplex S catheter along the long axis of the sciatic nerve behind the knee.
  Arms: LAX
Device: B Braun Contiplex S catheter

SUMMARY:
Displacement of popliteal sciatic nerve catheters after major foot and ankle surgery. A randomized controlled double blinded MRI study comparing long versus short axis catheter placement. Which procedure for insertion of nerve catheters for postoperative pain after major foot and ankle surgery is the best

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y.
* Major foot and ankle surgery postoperativ pain treatment with sciatic nerve catheter r
* Written and informed concent

Exclusion Criteria:

* Patient uanble to cooperate
* Patients not speaking and understanding Danish or English
* Patiens in immunosuppresive treatment
* Patienter with neuropathys in lower extremities
* Allergies to the in the protocole listes medicines
* A daily opoid intake
* Pregnant women
* Patients not meeting MR-criterias (metal, claustofobia...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Frequency of nerve catheter displacement | 48 hours after catheter placement

SECONDARY OUTCOMES:
Opioid comsumption | Within first 48 hours postoperatively
Number of rescue blocks | Within 48 hours postoperatively
Postoperativ pain after local anesthetic injection via sciatic nerve catheter | Within 48 hours postoperatively
MR evaluated distribution of local anesthetic after injection MR-contrast | 48 hours after catheter placement

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Aarhus University Hospital, Aarhus, Region Midt, Denmark

REFERENCES:
- [Background] di Benedetto P, Casati A, Bertini L, Fanelli G, Chelly JE. Postoperative analgesia with continuous sciatic nerve block after foot surgery: a prospective, randomized comparison between the popliteal and subgluteal approaches. Anesth Analg. 2002 Apr;94(4):996-1000, table of contents. doi: 10.1097/00000539-200204000-00041. PMID 11916811
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Tran DQ, Dugani S, Pham K, Al-Shaafi A, Finlayson RJ. A randomized comparison between subepineural and conventional ultrasound-guided popliteal sciatic nerve block. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):548-52. doi: 10.1097/AAP.0b013e318235f566. PMID 22005661
- [Background] Mariano ER, Kim TE, Funck N, Walters T, Wagner MJ, Harrison TK, Giori N, Woolson S, Ganaway T, Howard SK. A randomized comparison of long-and short-axis imaging for in-plane ultrasound-guided femoral perineural catheter insertion. J Ultrasound Med. 2013 Jan;32(1):149-56. doi: 10.7863/jum.2013.32.1.149. PMID 23269720
- [Background] Ironfield CM, Barrington MJ, Kluger R, Sites B. Are patients satisfied after peripheral nerve blockade? Results from an International Registry of Regional Anesthesia. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):48-55. doi: 10.1097/AAP.0000000000000038. PMID 24310051
- [Background] Marhofer D, Marhofer P, Triffterer L, Leonhardt M, Weber M, Zeitlinger M. Dislocation rates of perineural catheters: a volunteer study. Br J Anaesth. 2013 Nov;111(5):800-6. doi: 10.1093/bja/aet198. Epub 2013 Jun 7. PMID 23748198
- [Background] Niemi-Murola L, Krootila K, Kivisaari R, Kangasmaki A, Kivisaari L, Maunuksela EL. Localization of local anesthetic solution by magnetic resonance imaging. Ophthalmology. 2004 Feb;111(2):342-7. doi: 10.1016/j.ophtha.2003.05.026. PMID 15019387
- [Background] Compere V, Rey N, Baert O, Ouennich A, Fourdrinier V, Roussignol X, Beccari R, Dureuil B. Major complications after 400 continuous popliteal sciatic nerve blocks for post-operative analgesia. Acta Anaesthesiol Scand. 2009 Mar;53(3):339-45. doi: 10.1111/j.1399-6576.2008.01849.x. PMID 19243320
- [Background] Ilfeld BM, Sandhu NS, Loland VJ, Madison SJ, Suresh PJ, Mariano ER, Bishop ML, Schwartz AK, Lee DK. Ultrasound-guided (needle-in-plane) perineural catheter insertion: the effect of catheter-insertion distance on postoperative analgesia. Reg Anesth Pain Med. 2011 May-Jun;36(3):261-5. doi: 10.1097/AAP.0b013e31820f3b80. PMID 21519311
- [Background] Zacchino M, Almolla J, Canepari E, Merico V, Calliada F. Use of ultrasound-magnetic resonance image fusion to guide sacroiliac joint injections: a preliminary assessment. J Ultrasound. 2013 Jul 31;16(3):111-8. doi: 10.1007/s40477-013-0028-7. eCollection 2013 Jul 31. PMID 24432160
- [Derived] Hauritz RW, Pedersen EM, Linde FS, Kibak K, Borglum J, Bjoern S, Bendtsen TF. Displacement of popliteal sciatic nerve catheters after major foot and ankle surgery: a randomized controlled double-blinded magnetic resonance imaging study. Br J Anaesth. 2016 Aug;117(2):220-7. doi: 10.1093/bja/aew172. PMID 27440634